CLINICAL TRIAL: NCT03260621
Title: Cardiovascular Magnetic Resonance Real-time Exercise Stress Testing in Heart Failure With Preserved Ejection Fraction
Brief Title: CMR Exercise Stress Testing in HFpEF
Acronym: HFpEF-Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Andreas Schuster, PD Dr. med, University of Göttingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35/8/15
Record Dates: First submitted 2017-08-10; First posted 2017-08-24 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- echocardiographic increase in left atrial pressure (Other)
  Interventions: Diagnostic Test: stress CMR
- echocardiographic no increase in left atrial pressure (Other)
  Interventions: Diagnostic Test: stress CMR

INTERVENTIONS:
Diagnostic Test: stress CMR — additional stress CMR to the established clinical diagnostics

SUMMARY:
Patients of the University Hospital Göttingen with echocardiographic signs for diastolic heart failure and indication for right heart catheterisation will undergo additional diagnostic testing with CMR including exercise stress for detailed evaluation of diastolic dysfunction and tissue characterisation correlating the results with well-established clinical standards.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with dyspnoea under stress, echocardiographic criteria for diastolic dysfunction (E/E'>8) and clinical indication for right heart catheterisation

Exclusion Criteria:

* arrhythmia (brady- or tachycardic)
* bronchial asthma (allergic)
* incompliant patient
* pacemaker, ICD, non MRI-capable devices
* inability to use the ergometer in the MRI
* haemodynamic relevant valvular heart disease
* pulmonary disease (vital capacity or forced expiratory flow <80% of healthy control)
* angina pectoris
* post cardiac infarction
* anaemia (Hb <12 g/dl)
* uncontrollable hypertension (>150 mmHg systolic or >100 mmHg diastolic)
* age <18 years
* pregnancy
* claustrophobia
* renal insufficiency
* allergic to gadolinium based contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular magnetic resonance imaging | approx. 1 years
  ventricular and atrial volumes
Cardiovascular magnetic resonance imaging | approx. 1 years
  ventricular and atrial mechanics: strain
Cardiovascular magnetic resonance imaging | approx. 1 years
  quantification of extracellular volume (ECV)/interstitial fibrosis

OTHER OUTCOMES:
Exercise spirometry | approx. 1 years
  maximal oxygen uptake
Exercise spirometry | approx. 1 years
  respiratory quotient
Exercise spirometry | approx. 1 years
  power (watt/kg)
Right heart catheterization | approx. 1 years
  reference for intracardiac pressures: pulmonary artery pressure and pulmonary capillary wedge pressure

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schuster, MD, PhD, Principal Investigator — University of Göttingen
Locations (1):
- University Hospital Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data acquired within the current study will be available via the german centre for cardiovascular research (DZHK) to researchers who successfully applied to undertake additional scientific studies based on DZHK data.

REFERENCES:
- [Derived] Backhaus SJ, Schulz A, Lange T, Rosel SF, Schmidt-Schweda LS, Kutty S, Kowallick JT, Treiber J, Rolf A, Sossalla S, Hasenfuss G, Schuster A. Insights from serial cardiovascular magnetic resonance imaging show early progress in diastolic dysfunction relates to impaired right ventricular deformation. Sci Rep. 2025 Feb 3;15(1):4090. doi: 10.1038/s41598-025-87032-5. PMID 39900615
- [Derived] Schulz A, Schellinger IN, Backhaus SJ, Adler AS, Lange T, Evertz R, Kowallick JT, Hoffmann A, Matek C, Tsao PS, Hasenfuss G, Raaz U, Schuster A. Association of Cardiac MRI-derived Aortic Stiffness with Early Stages and Progression of Heart Failure with Preserved Ejection Fraction. Radiol Cardiothorac Imaging. 2024 Aug;6(4):e230344. doi: 10.1148/ryct.230344. PMID 39145733
- [Derived] Backhaus SJ, Nasopoulou A, Lange T, Schulz A, Evertz R, Kowallick JT, Hasenfuss G, Lamata P, Schuster A. Left Atrial Roof Enlargement Is a Distinct Feature of Heart Failure With Preserved Ejection Fraction. Circ Cardiovasc Imaging. 2024 Jul;17(7):e016424. doi: 10.1161/CIRCIMAGING.123.016424. Epub 2024 Jul 16. PMID 39012942
- [Derived] Backhaus SJ, Schulz A, Lange T, Evertz R, Kowallick JT, Hasenfuss G, Schuster A. Rest and exercise-stress estimated pulmonary capillary wedge pressure using real-time free-breathing cardiovascular magnetic resonance imaging. J Cardiovasc Magn Reson. 2024 Summer;26(1):101032. doi: 10.1016/j.jocmr.2024.101032. Epub 2024 Feb 29. PMID 38431079
- [Derived] Backhaus SJ, Schulz A, Lange T, Schmidt-Schweda LS, Evertz R, Kowallick J, Hasenfuss G, Schuster A. Real-time cardiovascular magnetic resonance imaging for non-invasive characterisation of heart failure with preserved ejection fraction: final outcomes of the HFpEF stress trial. Clin Res Cardiol. 2024 Mar;113(3):496-508. doi: 10.1007/s00392-023-02363-5. Epub 2024 Jan 3. PMID 38170248
- [Derived] Backhaus SJ, Lange T, Schulz A, Evertz R, Frey SM, Hasenfuss G, Schuster A. Cardiovascular magnetic resonance rest and exercise-stress left atrioventricular coupling index to detect diastolic dysfunction. Am J Physiol Heart Circ Physiol. 2023 May 1;324(5):H686-H695. doi: 10.1152/ajpheart.00081.2023. Epub 2023 Mar 10. PMID 36897745
- [Derived] Schuster A, Schulz A, Lange T, Evertz R, Hartmann F, Kowallick JT, Hellenkamp K, Uecker M, Seidler T, Hasenfuss G, Backhaus SJ. Concomitant latent pulmonary vascular disease leads to impaired global cardiac performance in heart failure with preserved ejection fraction. Eur J Heart Fail. 2023 Mar;25(3):322-331. doi: 10.1002/ejhf.2781. Epub 2023 Mar 2. PMID 36691723
- [Derived] Backhaus SJ, Uzun H, Rosel SF, Schulz A, Lange T, Crawley RJ, Evertz R, Hasenfuss G, Schuster A. Hemodynamic force assessment by cardiovascular magnetic resonance in HFpEF: A case-control substudy from the HFpEF stress trial. EBioMedicine. 2022 Dec;86:104334. doi: 10.1016/j.ebiom.2022.104334. Epub 2022 Nov 21. PMID 36423376
- [Derived] Backhaus SJ, Lange T, George EF, Hellenkamp K, Gertz RJ, Billing M, Wachter R, Steinmetz M, Kutty S, Raaz U, Lotz J, Friede T, Uecker M, Hasenfuss G, Seidler T, Schuster A. Exercise Stress Real-Time Cardiac Magnetic Resonance Imaging for Noninvasive Characterization of Heart Failure With Preserved Ejection Fraction: The HFpEF-Stress Trial. Circulation. 2021 Apr 13;143(15):1484-1498. doi: 10.1161/CIRCULATIONAHA.120.051542. Epub 2021 Jan 21. PMID 33472397